CLINICAL TRIAL: NCT02250846
Title: Phase II Study of EGFR-TKI in Patients With EGFR Mutation Non-Small Cell Lung Cancer With Asymptomatic Untreated Brain Metastasis
Brief Title: Study of EGFR-TKI to Asymptomatic Brain Metastases of NSCLC
Acronym: EABM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Gang Wu, cancer center, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WHXH-027
Record Dates: First submitted 2014-09-22; First posted 2014-09-26 (Estimated); Last update posted 2014-09-26 (Estimated); Status verified 2014-09

CONDITIONS: Asymptomatic Brain Metastases of Non Small Cell Lung Cancer
Keywords: EGFR mutations; asymptomatic brain metastases; EGFR-TKI; Erlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- arm a (Experimental): EGFR exon 19 mutation with EGFR-TKI
  Interventions: Drug: EGFR-TKI
- arm b (Experimental): EGFR exon 21 mutation with EGFR-TKI
  Interventions: Drug: EGFR-TKI

INTERVENTIONS:
Drug: EGFR-TKI — egfr-TKI treatment

SUMMARY:
The purpose of this study is to determine whether EGFR-TKI can control the development of intracranial lesions in Non Small Cell Lung Cancer patients with asymptomatic brain metastases, and the difference in progression free survival between exon 19 and exon 21 mutations.

DETAILED DESCRIPTION:
A open, positive control of phase II clinical trials, divided into selection period, treatment period and follow-up period , comply with the standard set of participants signed a written informed consent, according to different divided into 19 patients with EGFR mutations outside show son mutation group) and 21 extra show mutations, and according to the ECOG physical status, age, previous systemic treatments such as hierarchical analysis, regular follow-up and to assess efficacy, life care and safety.

ELIGIBILITY:
Inclusion Criteria:

1. at the age of 18 -70 years old, male or female
2. the non-small cell lung cancer diagnosed by histopathology
3. detected by ARMS to confirm that the EGFR sensitive mutant patients
4. the existence of MRI diagnosis of intracranial metastatic head enhancement, and the presence of imaging evaluating lesions (according to RECIST1.1)
5. have not received prior treatment of intracranial metastases, including radiotherapy, gamma knife, chemotherapy drugs
6. no brain metastasis symptoms, including, increased intracranial pressure, no vomiting, ignoring the papillary edema, no headache, without hemiplegia, ignore things not clear, without epilepsy
7. PS:0 or 1
8. the expected survival time 3 months >
9. patients signed informed consent voluntarily

Exclusion Criteria:

1. 4 weeks before entering the group received operation or operation, the wound has not healed completely
2. into group 2 weeks before receiving immune therapy or treatment of traditional Chinese Medicine
3. serious cardiovascular diseases, including Department of internal medicine, uncontrolled hypertension, unstable angina, myocardial infarction history exists within the past June, severe arrhythmia or pericardial effusion
4. serious infection, need intravenous antibiotic, antifungal or antiviral treatment
5. before entering the group 4 weeks participated in any study drug clinical trial
6. there are serious tumor invasion, oppression by the main bronchus or bronchial stenosis or obstruction, superior vena cava syndrome
7. the existence of herniation of brain tumor apoplexy, epilepsy, and frequent
8. suffering from a mental illness, poor compliance
9. the researchers think that do not fit into the group of cases

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2015-01; Primary Completion 2016-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Intracranial disease progression time | 20 months